CLINICAL TRIAL: NCT07264452
Title: Comparison of the Efficacy of Accelerated Intermittent Theta Burst Stimulation and Accelerated Continuous Theta Burst Stimulation in Patients With Treatment-Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Omer Faruk Uygur, associate professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-08/08; Atatürk University (Other: Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2025-11-21; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Treatment Resistant Depression (TRD); Transcranial Magnetic Stimulation; Accelerated Protocol; Intermittent Theta Burst Stimulation; Continuous Theta Burst Stimulation; Unilateral rTMS
Keywords: Treatment Resistant Depression (TRD); Transcranial Magnetic Stimulation; Accelerated protocol; intermittent theta burst stimulation; Continuous theta burst stimulation; Unilateral rTMS; unipolar major depressive disorder; non-invasive brain stimulation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itbs (Active Comparator): iTBS with eight digit coils to the left dorsolateral prefrontal cortex.
  Interventions: Device: Transcranial Magnetic Stimulation with figure-eight coil
- ctbs (Active Comparator): cTBS with a figure-of-eight coil to the right dorsolateral prefrontal cortex.
  Interventions: Device: Transcranial Magnetic Stimulation with figure-eight coil

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation with figure-eight coil — A total of 50 sessions will be administered to at least 30 patients, five sessions per day, five days a week for two weeks. There will be at least a 30-minute rest period between each session. One session for Group A involves a 5 Hz frequency intermittent theta burst stimulation (iTBS) protocol applied to the left DLPFC at 90-110% motor threshold.
  Other Names: A group
  Arms: Itbs
Device: Transcranial Magnetic Stimulation with figure-eight coil — The other patient group (Group B), consisting of at least 30 individuals, will receive 5 sessions per day, 5 days a week, for 2 weeks, for a total of 50 sessions. There will be at least a 30-minute rest period between each session. Group B will receive a 5 Hz, continuous theta burst stimulation (cTBS) protocol to the right DLPFC at 80% motor threshold.
  Other Names: B group
  Arms: ctbs

SUMMARY:
In recent years, research on the effectiveness of transcranial magnetic stimulation (TMS) in patients with treatment-resistant depression (RTD) has been steadily increasing. The aim of this study was to examine the effectiveness of accelerated unilateral application of two different forms of theta burst stimulation (TBU), a variation of repetitive TMU (rTMS)-intermittent TBU (iTBU) and continuous TBU (cTBU)-in TDD patients. The study aimed to compare the advantages of iTBU and cTBU protocols on depression, suicidal thoughts, anxiety levels, sleep disturbances, cognitive performance, and overall functioning following a two-week intensive treatment period and a 12-week follow-up period.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is the most common form of mood disorders that is frequently encountered in the society, has high recurrence and chronicity rates, and can lead to significant physical, cognitive, and psychosocial dysfunction in individuals. Although there is no single universally accepted definition for treatment-resistant depression (TRD), one of the most frequently used definitions is "failure to respond to at least two different antidepressant treatments for a sufficient duration and at an appropriate dose." Repetitive transcranial magnetic stimulation (rTMS) applied to the left and/or right dorsolateral prefrontal cortex (DLPFC) stands out as an alternative treatment approach in patients with TRD. One of these methods, theta-burst stimulation (TBS), is a non-invasive neuromodulation method approved by the US Food and Drug Administration (FDA) for treatment-resistant depression. Current methodological advances have enabled current TBS protocols to; Therapeutic efficacy can be enhanced by applying sessions multiple times a day, increasing the stimulation dose, and more precisely targeting the bilateral DLPFC. In addition to intermittent TBS (iTBS), continuous TBS (cTBS) protocols applied to the right DLPFC have also been reported to offer therapeutic potential in patients with TDD. Several studies have demonstrated that protocols consisting of 1,800 pulses produce lasting changes in cortical excitability and effectively trigger targeted neuroplastic mechanisms.

The study was planned to be conducted with patients who presented to the Atatürk University Faculty of Medicine, Department of Psychiatry Outpatient Clinic and were diagnosed with major depressive disorder (MDD) according to the American Psychiatric Association's DSM-5 diagnostic criteria. Participants were randomly assigned to two groups. In this single-blind, parallel study, one group was scheduled to receive a total of 50 sessions of iTBS to the left dorsolateral prefrontal cortex (left-DLPFC), while the other group received 50 sessions of cTBS to the right-DLPFC.

Clinical assessments of patients will be conducted at baseline, mid-treatment, at the end of treatment, and at weeks 2, 4, 8, and 12 post-treatment. Depressive symptoms will be measured with the HAM-D and MADRS, anxiety with the Hamilton Anxiety Rating Scale (HAM-A), sleep disturbances with the Pittsburgh Sleep Quality Index (PSQI) and Insomnia Severity Index (ISI), cognitive functions with the Montreal Cognitive Assessment Scale (MoCA), and functioning with the Brief Functioning Assessment Scale (BFAS). Participants were expected to maintain their current psychotropic medication at stable doses throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old
2. Patients diagnosed with Major Depressive Disorder according to DSM 5 and the severity of their illness
3. Scoring 7 points or more on the Maudsley staging method
4. Having depression unresponsive to 2 different antidepressants
5. No clinical mental retardation
6. Agree to participate in the study
7. Hamilton Depression Rating Scale-17 [HDRS] score of 20 or higher
8. Montgomery Asberg Depression Rating Scale [MADRS] score of 20 or above
9. Being right hand dominant
10. Having used the same antidepressant at the same dose for the last 4 weeks

Exclusion Criteria:

1. Diagnosed with a neurological or metabolic disease that affects cognitive functions (Systemic diseases such as diabetes mellitus, cardiovascular disease, cerebrovascular disease, chronic renal failure, Parkinson's disease, multiple sclerosis, polyneuropathy, inflammatory rheumatologic disease and malignancies)
2. Having a foreign body such as a pacemaker, intracranial implant that can magnetically interact
3. Hearing and visual impairments that prevent communication
4. Unstable or acute medical conditions
5. Pregnancy or breastfeeding
6. Having a primary psychiatric disorder other than major depressive disorder
7. Being diagnosed with severe MDD with psychotic features

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Depression severity | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  The Montgomery-Asberg Depression Rating Scale. The minimum and maximum scores are 0-60. Higher scores mean a worse outcome.
Depression severity | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  The Hamilton Depression Rating Scale-17. The minimum and maximum scores are 0-51. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Anxiety severity | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  Hamilton Anxiety Rating Scale. The minimum and maximum scores are 0-56. Higher scores mean a worse outcome.
Suicidal ideation score of The Hamilton Depression Rating Scale-17 | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  Suicidal ideation score on the third question of the Hamilton Depression Rating Scale-17. The minimum and maximum scores are 0-4. Higher scores mean a worse outcome.
Suicidal ideation score of The Montgomery-Asberg Depression Rating Scale | pretreatment, 1 week, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  Suicidal ideation score on the tenth question of the Montgomery-Asberg Depression Rating Scale. Minimum and maximum scores range from 0-6. Higher scores mean a worse outcome.
Insomnia Severity | pretreatment, 4 weeks, 10 weeks and 14 weeks
  It is measured with the Pittsburgh Sleep Quality Index (PSQI). The minimum and maximum scores are 0-21. Higher scores mean a worse outcome.
Insomnia Severity | pretreatment, 2 weeks, 4 weeks, 6 weeks, 10 weeks and 14 weeks
  It is measured with the Insomnia Severity Index (ISI). The minimum and maximum scores are 0-28. Higher scores mean a worse outcome.
Cognitive Assessment | pretreatment and 14 weeks
  Montreal Cognitive Assessment (MoCA) : The maximum score that can be obtained from the test is 30. A total score of 21 and above indicates that the participant is within normal limits.
Functionality Severity | pretreatment, 2 weeks and 14 weeks
  Functioning Assessment Short Test (FAST): It is used to measure patients' functionality. The minimum and maximum scores are 0-66. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Faruk UYGUR, Associate professor doctor, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No